CLINICAL TRIAL: NCT04073394
Title: "Mayo Clinic Diet" Individualized Lifestyle Intervention for Obesity Management Based on Obesity Phenotypes (PHENO-Diet Trial)
Brief Title: Individualized Lifestyle Intervention for Obesity Management Based on Obesity Phenotypes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Andres J. Acosta, M.D., Ph.D., Principal Investigator, Mayo Clinic
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-007485
Record Dates: First submitted 2019-08-28; First posted 2019-08-29 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2023-02

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Lifestyle Intervention (Active Comparator): Participants in this group will be instructed to follow a standard low calorie diet, recommended to have 30 minutes of physical activity 3-5 days per week, and will be followed by a wellness couch weekly.
  Interventions: Behavioral: Standard Lifestyle Intervention
- Modified Lifestyle Intervention (Experimental): Participants in this group will have a tailored diet, exercise, and behavioral plan according to their obesity phenotype.
  Interventions: Behavioral: Modified Lifestyle Intervention

INTERVENTIONS:
Behavioral: Standard Lifestyle Intervention — Research team will prescribe diet, exercise, behavioral plan for the participant to follow for the 12 week study. The lifestyle plan will be based on the Mayo Clinic Diet program.
  Arms: Standard Lifestyle Intervention
Behavioral: Modified Lifestyle Intervention — Research team will prescribe diet, exercise, behavioral plan for the participant to follow for the 12 week study. The lifestyle plan will be based on the participants obesity phenotype.
  Arms: Modified Lifestyle Intervention

SUMMARY:
The purpose of this protocol is to define an "individualized diet" approach based on obesity related phenotypes (pathophysiology obesity classification), which would increase weight loss, adherence, and weight loss maintenance.

ELIGIBILITY:
Inclusion Criteria:

* Adults with obesity (BMI >30Kg/m2); these will be otherwise healthy individuals with no unstable psychiatric disease and uncontrolled life-threatening comorbidities (i.e. unstable angina).
* Age: 18-65 years.
* Gender: Men or women.

Exclusion Criteria:

* Weight change greater than 3% in the previous 3 months (weight stable).
* History of bariatric surgery including lap band and bariatric endoscopy.
* Significant untreated psychiatric dysfunction including binge eating disorders and bulimia.
* Current use of anti-obesity pharmacotherapy, medications known to affect weight (e.g., corticosteroids) or GLP-1 agonist/analog for T2DM
* A positive score on the AUDIT-C questionnaire as judged by an investigator.
* Patient has a known history of any condition or factor judged by the investigator to preclude participation in the study or which might hinder study adherence

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 215 (Actual)
Dates: Start 2020-07-06 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
12-week total body weight loss | 12 weeks
  Change in body weight during the 12 week study

SECONDARY OUTCOMES:
Responder Rate | 12 weeks
  Proportion of patients losing > 3% of total body weight
Waist Circumference | 12 weeks
  Change in waist circumference (cm)
Fat Loss | 12 weeks
  Change in fat mass during the 12 week study using DEXA
Calorie Intake | 12 weeks
  Change in daily calorie intake
Calories to Fullness | 12 weeks
  Change in calories consumed to fullness during the 12 week study using satiation test
Gastric Emptying | 12 weeks
  Change in half gastric emptying time during the 12 week study using scintigraphy
Gastric Emptying 2 Hours | 12 weeks
  Change in gastric emptying percentage at 2 hours during the 12 week study using scintigraphy
Anxiety Level | 12 weeks
  Change is anxiety level during the 12 week study using the HADS-A scale
Emotional Eating | 12 weeks
  Change is emotional eating level during the 12 week study using the TFEQ score
Resting Metabolic Rate | 12 weeks
  Change in resting energy expenditure during the 12 week study using an indirect calorimetry
Adherence | 12 weeks
  Adherence and compliance with program defined by the number of contacts with the team

CONTACTS AND LOCATIONS:
Overall Officials: Andres Acosta, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Cifuentes L, Ghusn W, Feris F, Campos A, Sacoto D, De la Rosa A, McRae A, Rieck T, Mansfield S, Ewoldt J, Friend J, Grothe K, Lennon RJ, Hurtado MD, Clark MM, Camilleri M, Hensrud DD, Acosta A. Phenotype tailored lifestyle intervention on weight loss and cardiometabolic risk factors in adults with obesity: a single-centre, non-randomised, proof-of-concept study. EClinicalMedicine. 2023 Mar 24;58:101923. doi: 10.1016/j.eclinm.2023.101923. eCollection 2023 Apr. PMID 37007741
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials